CLINICAL TRIAL: NCT05086328
Title: The Effect of Nonviolent Resistance in Parent Group Training in Child Psychiatric Care
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: 2021 GV OUG
Record Dates: First submitted 2021-08-31; First posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Helplessness, Learned; Family Conflict; Mentalising; Parenting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Nonviolent Resistance — Six two weekly sessions of two hours, based on nonviolent resistance Questionnaires pre and post intervention

SUMMARY:
In a Flemish sample of parents of children with psychiatric problems, this study evaluates the effect of a parent group training based on nonviolent resistance on family functioning, parenting variables and mental states of the parents, pre- and post-training.

DETAILED DESCRIPTION:
Nonviolent Resistance (NVR) is an intervention method for families and teams that are suffering from helplessness and hopelessness. By empowering individuals through specific focus points and techniques, they can re-establish their role as authority figures for the child. The child, exhibiting dangerous and/or coercive behavior, can feel reconnected and guided.

Previous research has shown that parents score higher on General family functioning, Affective reactions and affective involvement, and Role definitions, but not Behavioral control, Problem solving and Communication. Positive effects were visible at a follow up moment, three months later. Parents reported significantly lower on anxiety for the aggression of their child, the self-efficiency about parental capacities and received social support. General parenting stress diminished significantly. A control group showed no such significant changes.

Participants with specific problems and waiting to be admitted in the residential ward at the study location can receive pre-care, in the form of a parental group training based on NVR. In six two weekly sessions, combined with intermediate telephone support and home assignments, parents are involved in important parent-child-oriented aspects.

This study will evaluate the effect of the training in a Flemish sample, focusing on family functioning, parenting variables and reflective functioning of the parents, pre- and post-training. T1 is at the time between invitation to participate and the first session; T2 is in the first week after the last session (T1 + 12 to 14 weeks); T3 is at three months after the last session; T4 is at six months after the last session.

The following primary outcomes are expected after the parent group:

* More behavior and mental states pointing towards NVR
* More use of adequate emotion regulation
* Less behavioral problems in the child

Secondary outcomes are expected, according to previous research measuring indirect effects of NVR treatment

* More adequate attunement to child
* More cohesion and structure in the family
* More adequate parenting behavior
* Less stress and burdening for parents

The investigators also expect parents with a more secure attachment style to benefit more (T2) and longer (T3 and T4) from the training.

ELIGIBILITY:
Inclusion Criteria:

Parents engage in the NVR training of the child psychiatric clinic at the study location for at least 5 out of 6 training sessions

Exclusion Criteria:

* insufficient understanding of Dutch/Flemish language
* simultaneously following a different parent group treatment, external to the study location

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: - parents of child on the waiting list or already admitted for help in the child psychiatric clinic at the study location, with specific parental stress related to helplessness
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline mean scores in four domains of Nonviolent Resistance as measured with the Parental Anchoring Scale (Flemish version) | T1 baseline = 1 to 2 weeks before first session; T2 = T1 + 12 to 14 weeks; T3 = T2 + three months; T4 = T2 + six months
  The Parental Anchoring Questionnaire (Flemish version = OAFS) measures Presence, Self-Control, Social Support, and Structure, on a 7-point scale. High scores mean more Nonviolent Resistance.
Change from baseline mean scores in child behavior as measured with the Child Behavior Checklist (CBCL) | T1 baseline = 1 to 2 weeks before first session; T2 = T1 + 12 to 14 weeks; T3 = T2 + three months; T4 = T2 + six months
  The CBCL is a general questionnaire measuring internalizing and externalizing behavior of the child as perceived by the parents, using a 3-point scale. High scores mean more problems.
Change from baseline mean scores in emotion regulation as measured with the Emotion Regulation Questionnaire (ERQ) | T1 baseline = 1 to 2 weeks before first session; T2 = T1 + 12 to 14 weeks; T3 = T2 + three months; T4 = T2 + six months
  The ERQ measures Reappraisal and Suppression as two distinct mechanisms to deal with emotional problems. Reappraisal is related more with healthy coping. A 7-point scale leads to scores pointing to high Reappraisal and high Suppression.

SECONDARY OUTCOMES:
Change from baseline mean scores in attunement to the child as measured with the Parental Reflective Functioning Scale (PRFQ) | T1 baseline = 1 to 2 weeks before first session; T2 = T1 + 12 to 14 weeks; T3 = T2 + three months; T4 = T2 + six months
  The PRFQ measures reflective functioning or mentalizing, a process essential in developing a secure attachment and positive attunement to the child. There are three subscales with a 7-point scale: Pre-mentalizing (PM), Certainty about Mental States (CMS), and Interest and Curiosity in Mental States (IC).
Change from baseline mean scores in family functioning as measured with the Questionnaire for Family Functioning (VGFO) | T1 baseline = 1 to 2 weeks before first session; T2 = T1 + 12 to 14 weeks; T3 = T2 + three months; T4 = T2 + six months
  The VGFO measures Basic care, Education, Social contacts, Youth experiences (of parents), and the Partner relationship, each on a 5-point scale.
Change from baseline mean scores in parental burden as measured with the Parental Burden Questionnaire (OBVL) | T1 baseline = 1 to 2 weeks before first session; T2 = T1 + 12 to 14 weeks; T3 = T2 + three months; T4 = T2 + six months
  The OBVL measures possible sources of burden for parents in five scales: Parent-child relationship, Parenting competency, Depressed mood (of the parent), Role restriction, Health complaints, all on a 4-point scale. Higher scores mean more burden for the parents.
Change from baseline mean scores in parental behavior as measured with the Short Scale for Parental Behavior (VSOG) | T1 baseline = 1 to 2 weeks before first session; T2 = T1 + 12 to 14 weeks; T3 = T2 + three months; T4 = T2 + six months
  The VSOG measures five different types of parental behavior on a 5-point scale: Positive engagement, Setting/teaching rules, Material rewarding, Punishing, and Physical punishment.

CONTACTS AND LOCATIONS:
Overall Officials: Bart Colson, MA, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sherman, E. (2018). Group-Based Nonviolent Resistance Program: Development of a Short-Term Intervention and Preliminary Assessment of Its Feasibility and Acceptance. Tel Aviv University, Master Thesis
- [Background] Omer H, Lebowitz ER. Nonviolent Resistance: Helping Caregivers Reduce Problematic Behaviors in Children and Adolescents. J Marital Fam Ther. 2016 Oct;42(4):688-700. doi: 10.1111/jmft.12168. Epub 2016 Jun 13. PMID 27292182
- [Result] Kiliçarslan, S. (2019). The Effect of the Non-violent Resistance Program for the Parents of Children with Violent Behaviors. Kastamonu Education, 27(2), 701-716. https://doi.org/10.24106/kefdergi.2691
- [Result] Kiliçarslani, S., Ördem, S., Taltekin, A. & Ardiç, R. (2019). The Effect of Non-Violent Resistance Program on Family Relationships and Parentship Perceptions of Parents. PAU Journal of Education, 45, 211-234. doi: 10.9779/PUJE.2018.230
- [Result] Schorr-Sapir I, Gershy N, Apter A, Omer H. Parent training in non-violent resistance for children with attention deficit hyperactivity disorder: a controlled outcome study. Eur Child Adolesc Psychiatry. 2022 Jun;31(6):929-938. doi: 10.1007/s00787-021-01723-8. Epub 2021 Feb 2. PMID 33528659
- [Result] Van Holen F, Vanderfaeillie J, Omer H. Adaptation and Evaluation of a Nonviolent Resistance Intervention for Foster Parents: A Progress Report. J Marital Fam Ther. 2016 Apr;42(2):256-71. doi: 10.1111/jmft.12125. Epub 2015 Apr 24. PMID 25907660